CLINICAL TRIAL: NCT00415194
Title: A Randomized Phase 3 Study of Pemetrexed in Combination With Cisplatin Versus Cisplatin Monotherapy in Patients With Recurrent or Metastatic Head and Neck Cancer
Brief Title: A Study for Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8431; H3E-MC-JMHR (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Results first posted 2011-04-06 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pemetrexed/Cisplatin (Experimental): Pemetrexed 500 milligrams per meter square (mg/m^2) administered intravenously (IV) plus cisplatin 75 mg/m^2 IV on Day 1 every 21 days. Pretreatment, Both Treatment Arms: Dexamethasone administered orally (po): 4 milligrams (mg) twice daily (BID) taken on the day before, the day of, and day after study treatment.
  Vitamin B12 administered intramuscularly (im): 1000 micrograms (μg) taken 1 to 2 weeks before treatment and every 9 weeks until 3 weeks after last treatment dose. Folic Acid administered orally (po): 350 μg to 1000 μg taken 1 to 2 weeks before treatment and continue daily until 3 weeks after last treatment dose.
  Interventions: Drug: pemetrexed; Drug: cisplatin
- Placebo/Cisplatin (Placebo Comparator): Placebo (approximately 100 mL normal saline) administered intravenously (IV) plus cisplatin 75 mg/m^2 on Day 1 every 21 days.
  Pretreatment - Both Treatment Arms: Dexamethasone administered orally (po): 4 milligrams (mg) twice daily (BID) taken on the day before, the day of, and day after study treatment. Vitamin B12 administered intramuscularly (im): 1000 micrograms (μg) taken 1 to 2 weeks before treatment and every 9 weeks until 3 weeks after last treatment dose.
  Folic Acid administered orally (po): 350 μg to 1000 μg taken 1 to 2 weeks before treatment and continue daily until 3 weeks after last treatment dose.
  Interventions: Drug: cisplatin; Drug: placebo

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m^2, IV, every 21 days, six 21 day cycles
  Other Names: Alimta; LY231514
  Arms: Pemetrexed/Cisplatin
Drug: cisplatin — 75 mg/m^2, administered IV, every 21 days, six 21 day cycles
Drug: placebo — Approximately 100 mL normal saline administered IV, every 21 days, six 21 day cycles
  Arms: Placebo/Cisplatin

SUMMARY:
This study will compare the effects of pemetrexed plus cisplatin versus cisplatin alone in head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* You must have head and neck cancer that has returned and cannot be treated with surgery or other types of treatment. OR You must have head and neck cancer that was just found and has spread to other parts of your body.
* You must have a performance status of 0,1 or 2. This means that you must at least be able to get around, be able to take care of yourself and must be up and about most of the day.
* Your test results must show that your liver, kidneys and blood cells are working normally.
* You must understand and sign the form that gives your agreement to willingly be part of the study.
* You must be at least 18 years of age.

Exclusion Criteria:

* You cannot have previously been given other treatment for cancer that has spread to other parts of your body.
* You cannot have a serious sickness that might keep you from finishing the study (for example a bad infection).
* You cannot have any extra fluid in your chest or bowel area unless your doctor tells you it can be drained before you join the study.
* You cannot have any cancer called nasopharyngeal cancer, paranasal sinus cancer, lip cancer, or salivary gland cancer.
* If you are taking high dose aspirin or other medicines called non-steroidal anti-inflammatory drugs and cannot stop taking them for at least 5 days, you cannot be in the study. Your doctor or a member of the study team can explain which drugs are non-steroidal anti-inflammatory drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (94):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beech Grove, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stony Brook, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Smithfield, Rhode Island
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., S.M. de Tucuman
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Fé
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucumain
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belo Horizonte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
- China (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanning
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odense
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avignon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- Germany (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
- India (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bhopal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolkata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Patna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Confreria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
- Mexico (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durango
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Michoacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma Sur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toluca
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnaul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelyabinsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Murmansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parktown
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hwasun-Gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Murcia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hualien City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liouying/Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed/Cisplatin: Pemetrexed 500 milligrams per meter square (mg/m^2) administered intravenously (IV) plus cisplatin 75 mg/m^2 IV on Day 1 every 21 days.
  Pretreatment - Both Treatment Arms: Dexamethasone administered orally (po): 4 milligrams (mg) twice daily (BID) taken on the day before, the day of, and day after study treatment.
  Vitamin B12 administered intramuscularly (im): 1000 micrograms (μg) taken 1 to 2 weeks before treatment and every 9 weeks until 3 weeks after last treatment dose.
  Folic Acid administered orally (po): 350 μg to 1000 μg taken 1 to 2 weeks before treatment and continue daily until 3 weeks after last treatment dose.
- Placebo/Cisplatin: Placebo (approximately 100 mL normal saline) administered IV plus cisplatin 75 mg/m^2 on Day 1 every 21 days.
  Pretreatment - Both Treatment Arms: Dexamethasone administered orally (po): 4 milligrams (mg) twice daily (BID) taken on the day before, the day of, and day after study treatment.
  Vitamin B12 administered intramuscularly (im): 1000 micrograms (μg) taken 1 to 2 weeks before treatment and every 9 weeks until 3 weeks after last treatment dose.
  Folic Acid administered orally (po): 350 μg to 1000 μg taken 1 to 2 weeks before treatment and continue daily until 3 weeks after last treatment dose.
Period: Overall Study
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin
Started | 398 | 397
Received at Least 1 Dose of Study Drug | 392 | 385
Completed | 70 | 55
Not Completed | 328 | 342
Not completed — Adverse Event | 37 | 32
Not completed — Entry Criteria Not Met | 4 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 10 | 16
Not completed — Progressive Disease | 180 | 217
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 28 | 21
Not completed — Death Due to Study Disease | 26 | 29
Not completed — Death Due to Study Drug Related AE | 11 | 1
Not completed — Death Due to Procedural Related AE | 0 | 1
Not completed — Death Due to AE (Other Causes) | 27 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin | Total
Number analyzed (Participants) | 398 | 397 | 795
Age Continuous [Mean (Standard Deviation); unit: years] | 57.45 (9.54) | 57.78 (9.36) | 57.62 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 53 | 109
  Male | 342 | 344 | 686
Race/Ethnicity, Customized [Number; unit: Participants]
  African | 17 | 12 | 29
  Caucasian | 243 | 233 | 476
  East Asian | 55 | 65 | 120
  Hispanic | 11 | 16 | 27
  West Asian (Indian sub-continent) | 72 | 70 | 142
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Argentina | 5 | 10 | 15
  Belgium | 7 | 10 | 17
  Brazil | 16 | 12 | 28
  China | 5 | 7 | 12
  Denmark | 7 | 3 | 10
  France | 3 | 3 | 6
  Germany | 50 | 48 | 98
  Hungary | 23 | 22 | 45
  India | 72 | 75 | 147
  Italy | 19 | 21 | 40
  Korea, Republic of | 29 | 24 | 53
  Mexico | 9 | 8 | 17
  Netherlands | 8 | 11 | 19
  Poland | 10 | 10 | 20
  Romania | 20 | 22 | 42
  Russian Federation | 23 | 20 | 43
  South Africa | 11 | 9 | 20
  Spain | 31 | 29 | 60
  Taiwan | 21 | 25 | 46
  United States | 29 | 28 | 57
Previously Treated for Head and Neck Cancer (HNC) [Number; unit: Participants]
  No | 35 | 39 | 74
  Yes | 363 | 358 | 721
Prior Treatment with Platinum-Based Therapy [Number; unit: Participants]
  No | 213 | 228 | 441
  Yes | 185 | 169 | 354
Distant Metastasis [Number; unit: Participants]
  No | 165 | 155 | 320
  Yes | 233 | 242 | 475
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — These scales and criteria are used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis:
  1. Fully active, able to carry on all pre-disease performance without restriction
  2. Restricted in strenuous activity,able to carry out work of a light or sedentary nature
  3. Ambulatory, but unable to carry out any work activities. Capable of only limited selfcare
  4. Completely disabled. Cannot carry on any selfcare.
  5. Dead
  Participants
    0 | 90 | 90 | 180
    1 | 257 | 253 | 510
    2 | 51 | 53 | 104
    Missing Data | 0 | 1 | 1
Primary Site of Disease [Number; unit: Participants]
  Hypopharynx | 63 | 59 | 122
  Larynx | 103 | 102 | 205
  Oral Cavity | 138 | 123 | 261
  Oropharynx | 86 | 106 | 192
  Other | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS duration is defined as the time from the date of randomization to the date of death from any cause. For each participant who is not known to have died as of the data-inclusion cut-off date, OS duration will be censored at the date of the participant's last contact prior to that cut-off date.
Time Frame: Baseline to date of death from any cause up to 36 months
Population: Intention to Treat (ITT) Population - defines the treatment group as those to which participants were assigned by random allocation, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin
Number analyzed (Participants) | 398 | 397
Months | 7.33 [6.34 to 8.38] | 6.28 [5.52 to 7.06]
Statistical Analysis 1: Comparison: Pemetrexed/Cisplatin vs Placebo/Cisplatin; Test type: Superiority or Other; p = 0.082, Stratified Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.75 to 1.02]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Objective PFS is defined as the time from date of randomization to date of objectively determined progressive disease (PD) or death from any cause, whichever comes first. PD was defined by Response Evaluation Criteria in Solid Tumors (RECIST). PD=at least a 20% increase in sum of longest diameter of target lesions. For participants who are not known to have died as of the data-inclusion cut-off date, and who do not have progressive disease, PFS will be censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systemic anticancer therapy.
Time Frame: baseline to measured progressive disease up to 33 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin
Number analyzed (Participants) | 398 | 397
months | 3.61 [3.15 to 4.07] | 2.79 [2.69 to 3.22]
Statistical Analysis 1: Comparison: Pemetrexed/Cisplatin vs Placebo/Cisplatin; Test type: Superiority or Other; p = 0.166, Stratified Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.76 to 1.03]

3. Secondary Outcome: Percent of Participants With a Tumor Response (Response Rate)
Description: Tumor Response is evaluated as CR (Complete Response) or PR (Partial Response) per Response Evaluation Criteria in Solid Tumors (RECIST criteria). Possible evaluations include: CR: Disappearance of all target lesions. PR: At least a 30% decrease in the size of target lesions. Response rate (%) = (number of participants with CR+PR/number of participants)*100
Time Frame: Baseline to progressive disease or discontinuation of study treatment up to 11 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin
Number analyzed (Participants) | 398 | 397
Percentage of participants | 12.1 | 8.1
Statistical Analysis 1: Comparison: Pemetrexed/Cisplatin vs Placebo/Cisplatin; Test type: Superiority or Other; p = 0.061, Unadjusted normal distribution; p-value is based on an unadjusted, normal distribution approximation for differences in rates

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR is time from first observation of complete response (CR) or partial response (PR) to first observation of PD or death. Response is objective status of CR or PR using RECIST criteria. CR is disappearance of lesions. PR is >30% decrease in size of lesions. Responder is any participant with CR or PR. PD is at least 20% increase in sum of longest diameter of target lesions. For participants alive as of data-inclusion cut-off date and who do not have PD, DoR will be censored at date of last objective progression-free disease assessment before date of any subsequent systemic anticancer therapy.
Time Frame: time of response to progressive disease up to 24 months
Population: ITT population with a confirmed best response of complete response (CR) or partial response (PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin
Number analyzed (Participants) | 48 | 32
Months | 5.29 [4.21 to 5.98] | 4.37 [3.58 to 6.44]
Statistical Analysis 1: Comparison: Pemetrexed/Cisplatin vs Placebo/Cisplatin; Test type: Superiority or Other; p = 0.811, Stratified Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.56 to 1.53]

5. Secondary Outcome: Time to Treatment Worsening in Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N) Total Score
Description: FACT-H&N consists of 39 items with 5-point rating scale from 0 (not at all) to 4 (very much). FACT-H&N Total score ranges from 0 to 148. Higher score represents a better quality of life. Time to worsening was defined as the first date of worsening in the FACT H&N Total score that was considered at least the prospectively defined minimally important difference (MID) as compared with participant's baseline score, or date of death from any cause. The MID for FACT H&N Total score was a decrease of 12 points.
Time Frame: Baseline (</=Day 1 of first dose) and Day 1 of every subsequent cycle to 30-day post-study completion up to 33 months
Population: Intention to treat (ITT) population with at least Baseline data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin
Number analyzed (Participants) | 271 | 270
Months | 3.29 [2.76 to 4.11] | 2.89 [2.40 to 3.19]
Statistical Analysis 1: Comparison: Pemetrexed/Cisplatin vs Placebo/Cisplatin; Test type: Superiority or Other; p = 0.20, Stratified Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.69 to 1.07]

6. Secondary Outcome: Correlation Between Biomarkers and Treatment Effect
Description: Correlation between highly up/downregulated genes and clinical response (Overall Survival (OS) and Progression-Free Survival (PFS)). OS is is defined as the time from the date of randomization to the date of death from any cause. PFS is defined as the time from the date of randomization to the date of objectively determined progressive disease or death from any cause, whichever comes first.
  0 participants were analyzed; Reason: The relatively low number of samples collected would not have yielded a meaningful genomic analysis and the decision was made to not analyze the data.
Time Frame: Baseline
Population: Zero participants were analyzed because the relatively low number of samples collected would not have yielded a meaningful genomic analysis.
Measure: Number; unit: correlation coefficient
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Participants who received at least one dose of study drug were included in the safety population included here.
Groups:
- Pemetrexed/Cisplatin: Pemetrexed 500 milligrams per meter square (mg/m2) administered intravenously (IV) plus cisplatin 75 mg/m2 IV on Day 1 every 21 days. Pretreatment - Both Treatment Arms: Dexamethasone administered orally (po): 4 milligrams (mg) twice daily (BID) taken on the day before, the day of, and day after study treatment. Vitamin B12 administered intramuscularly (im): 1000 micrograms (μg) taken 1 to 2 weeks before treatment and every 9 weeks until 3 weeks after last treatment dose. Folic Acid administered orally (po): 350 μg to 1000 μg taken 1 to 2 weeks before treatment and continue daily until 3 weeks after last treatment dose.
- Placebo/Cisplatin: Placebo (approximately 100 mL normal saline) administered IV plus cisplatin 75 mg/m2 on Day 1 every 21 days. Pretreatment - Both Treatment Arms: Dexamethasone administered orally (po): 4 milligrams (mg) twice daily (BID) taken on the day before, the day of, and day after study treatment. Vitamin B12 administered intramuscularly (im): 1000 micrograms (μg) taken 1 to 2 weeks before treatment and every 9 weeks until 3 weeks after last treatment dose. Folic Acid administered orally (po): 350 μg to 1000 μg taken 1 to 2 weeks before treatment and continue daily until 3 weeks after last treatment dose.
Arm/Group | Pemetrexed/Cisplatin | Placebo/Cisplatin
Serious Adverse Events (participants affected / at risk) | 185/392 | 132/385
Other Adverse Events (participants affected / at risk) | 343/392 | 316/385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Cisplatin (N=392) | Placebo/Cisplatin (N=385)
Agranulocytosis (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 22 (27) | 17 (20)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow toxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (13) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 14 (16) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 12 (13) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (12) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 1 (1)
Aphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 1 (1)
Disbacteriosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 3 (3)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 13 (14) | 7 (7)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (24) | 9 (9)
Adhesion (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 6 (8) | 9 (9)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 4 (4) | 4 (4)
Face oedema (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 7 (7) | 5 (5)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Performance status decreased (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 9 (9) | 6 (7)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acinetobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Central line infection (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 26 (29) | 7 (9)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 4 (4)
Septic shock (Infections and infestations) | 3 (3) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 3 (3)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspiration bronchial (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 1 (1)
Blood electrolytes abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 2 (2)
ECG signs of myocardial ischaemia (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 7 (9) | 4 (4)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 5 (6)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 9 (9) | 7 (7)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Hypophagia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (6)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (4) | 4 (4)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 7 (9) | 4 (5)
Renal failure acute (Renal and urinary disorders) | 3 (4) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 15 (15)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 4 (4) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena caval occlusion (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Cisplatin (N=392) | Placebo/Cisplatin (N=385)
Anaemia (Blood and lymphatic system disorders) | 118 (133) | 79 (88)
Leukopenia (Blood and lymphatic system disorders) | 38 (57) | 24 (35)
Neutropenia (Blood and lymphatic system disorders) | 67 (105) | 35 (48)
Thrombocytopenia (Blood and lymphatic system disorders) | 28 (33) | 17 (22)
Constipation (Gastrointestinal disorders) | 56 (63) | 53 (65)
Diarrhoea (Gastrointestinal disorders) | 42 (50) | 33 (35)
Dysphagia (Gastrointestinal disorders) | 19 (19) | 22 (23)
Nausea (Gastrointestinal disorders) | 118 (199) | 106 (153)
Vomiting (Gastrointestinal disorders) | 62 (81) | 79 (104)
Asthenia (General disorders) | 36 (41) | 31 (35)
Fatigue (General disorders) | 67 (88) | 53 (57)
Mucosal inflammation (General disorders) | 25 (30) | 8 (8)
Pain (General disorders) | 16 (19) | 20 (23)
Pyrexia (General disorders) | 40 (44) | 19 (21)
Creatinine renal clearance decreased (Investigations) | 32 (34) | 31 (36)
Weight decreased (Investigations) | 45 (47) | 50 (51)
Anorexia (Metabolism and nutrition disorders) | 52 (63) | 44 (50)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (28) | 14 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 40 (47) | 29 (30)
Hyponatraemia (Metabolism and nutrition disorders) | 21 (27) | 24 (25)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (25) | 23 (26)
Insomnia (Psychiatric disorders) | 23 (24) | 23 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 20 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days